CLINICAL TRIAL: NCT02841878
Title: Genetic Determinism of Epithelial Barrier Defects Induced by Increase in Proteases Activity in Irritable Bowel Syndrome
Brief Title: Genetic Determinism of Epithelial Barrier Defects in Irritable Bowel Syndrome
Acronym: PROTIBS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Decision of the investigator
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 14-PP-20
Record Dates: First submitted 2015-08-24; First posted 2016-07-22 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Irritable Bowel Syndrome (IBS)
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- analysis on colorectal biopsy (Other): * Proteases activity (cystein and serin proteases)
  * Proteases inhibitors genes expression (Serpins A1 / E1)
  * Colonic biopsies permeabilityTight junctions genes expression
  * Cytokines genes expression (TNFalpha, interleukines)
  * Cellularity on histologic sections
  Interventions: Genetic: Analysis on colorectal biopsy

INTERVENTIONS:
Genetic: Analysis on colorectal biopsy

SUMMARY:
Irritable bowel syndrome (IBS) profoundly affects the quality of life. Mucosal micro-inflammation, epithelial permeability disorder and proteases activity increase have been demonstrated in the patients' gastrointestinal tract. Protease activity increase could be subjected to a genetic determinism (decrease in proteases inhibitors genes expression). Objectives: 1/ To study relations between proteases activity (in stool and colonic biopsies supernatants), proteases inhibitors genes expression and mucosal cellular infiltrate (IBS patients and healthy subjects). 2/ Establishing a correlation between proteases activity, mucosal micro-inflammation and symptoms. 3/ To evaluate proteases inhibitors therapeutic potential. Expected results: 1/ Decreased expression of proteases inhibitors genes in subjects with IBS. 2/ Correlation of symptoms with proteases activity intensity. 3/ Demonstration of restorative potential of proteases inhibitors.

DETAILED DESCRIPTION:
Irritable bowel syndrome (IBS) is the first reason for consultation in gastroenterology and his prevalence reach 5% of the general population. IBS is characterized by abdominal discomfort, diarrhea or constipation and decreased quality of life.

Recent facts on IBS pathophysiology show association between mucosal immunity activation (mast cells and their proteases) and epithelial permeability disorder. Permeability disorder can be reproduced by application of colonic biopsies cultures supernatants on in-vitro cell cultures. In parallel, tight junctions proteins mRNA (ZO-1, Occludin) decrease is observed ex-vivo in biopsies and in-vitro.

Gut bacterial proteases (cystein and serin proteases) may also play a role. In human, proteases activity is correlated with IBS symptoms severity. Proteases activity increase (cystein and serin proteases) is poorly understood, and this increase could be subjected to a genetic determinism (decrease in proteases inhibitors genes expression - Serpin A1/E1).

Objectives: 1/ To study relations between proteases activity (in stool and colonic biopsies supernatants), proteases inhibitors genes expression and mucosal cellular infiltrate (IBS patients and healthy subjects). 2/ Establishing a correlation between proteases activity, mucosal micro-inflammation and symptoms. 3/ To evaluate proteases inhibitors therapeutic potential.

Method: Subjects will be recruited in gastroenterology consultation. IBS patients will answer to Rome III criteria. Patients coming for screening colonoscopy will be defined as healthy subjects.

Colonic biopsies will be sent in real time to the research laboratory (EA 6302) for supernatants collecting, mRNA expression studies (Serpins, ZO-1, occludin, cytokines), proteases activity / permeability measurements and proteases inhibitors reversibility tests. Histologic study will also be performed.

Expected results: 1/ Decreased expression of proteases inhibitors genes in subjects with IBS. 2/ Correlation of symptoms with proteases activity intensity. 3/ Demonstration of restorative potential of proteases inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* Patient with irritable bowel syndrome (IBS), defined by Rome III criteria (patient group)
* Patients coming for screening colonoscopy (control group)

Patients exclusion criteria :

* Active inflammatory bowel disease
* Infectious bowel disease or other cause that could explain digestive symptoms

Healthy subjects inclusion criteria :

* Patients coming for screening colonoscopy without inflammatory bowel disease or IBS

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-09 (Estimated); Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Clinical criteria | at the medical visit
  Abdominal Pain : Francis scoring
Clinical criteria | at day one
  Transit disorders : Rome III criteria questionnaire
Clinical criteria | at day one
  Quality of life alteration (questionnaires)

SECONDARY OUTCOMES:
Experimental criteria | at day one
  Proteases activity (cystein and serin proteases)
  Tight junctions genes expression Cytokines genes expression (TNFalpha, interleukines) Cellularity on histologic sections
Experimental criteria | at day one
  Proteases inhibitors genes expression (Serpins A1 / E1)
Experimental criteria | at day one
  Colonic biopsies permeability

CONTACTS AND LOCATIONS:
Overall Officials: Thierry PICHE, MD, Principal Investigator — Nice University Hospital
Locations (1):
- Department of gastroenterology, Hopital Archet 2, Nice, France